CLINICAL TRIAL: NCT03314272
Title: Automated Versus Conventional Perioperative Glycemic Control in Adult Diabetic Patients Undergoing Cardiopulmonary Bypass Surgery
Brief Title: Automated vs Conventional Perioperative Glycemic Control in Diabetic Patients Undergoing Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Roland Kaddoum, Associate Professor Department of Anesthesiology/ Director of Pediatric Anesthesia/ Director of Operating Room, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES.RK.03
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Diabetes; Cardiopulmonary Bypass
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sliding scale protocol (No Intervention): Consists of giving insulin every 30 minutes based on the blood glucose readings as follows:
  * <150 mg/dl: 0 units of insulin
  * 150-220 mg/dl: 2 units of insulin
  * 201-250 mg/dl: 4 units
  * 251-300 mg/dl: 6 units
  * 301-350 mg/dl: 8 units
  * 351-400 mg/dl: 10 units
  * > 400 mg/dl: inform the MD on call
- Space Glucose Control (Experimental): Automated protocol consisting of an insulin infusion pump named The Space Glucose Control System.
  Intervention:
  For glucose measurement, a sample of blood gas will be taken every 30 minutes. Actrapid HM will be used in a 4IU/ ml concentration for infusion in a 50 ml syringe.
  The range of glucose will be recorded throughout the intra-operative period. The number of hypoglycemic (<70mg/dl) and hyperglycemic (> 200mg/dl) events will be recorded.
  Interventions: Device: Space Glucose Control

INTERVENTIONS:
Device: Space Glucose Control — Development of a closed loop control system via Space Glucose Control that automatically infuses insulin on the basis of an automated algorithm, which integrates a continuous glucose signal, could help overcome these obstacles and permit strict glycemic control without increasing the workload.
  Arms: Space Glucose Control

SUMMARY:
The purpose of this randomized controlled trial is to evaluate a fully automated algorithm for the establishment of glycemic control in diabetic patients and to compare the results with routine management of hyperglycemia in patients undergoing cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
Upon admission of the patients to the hospital, demographic and physiological data will be collected including waist circumference and BMI. A set of baseline laboratory tests will be done for each patient including: glucose level, Hba1c, lipid profile, creatinine level, liver enzymes and micro albumin/creatinine urinary ratio.

Patients will be asked about the presence of any diabetes complications: nephropathy, retinopathy and/or neuropathy.

In the induction room, an intravenous cannula will be inserted by an experienced anesthesiology staff or resident. A three way stopcock will be connected directly to the cannula. Standard monitors (ECG, non-invasive blood pressure and oxygen saturation) will be connected to the patient. An arterial line will be inserted by the anesthesia resident under sterile conditions using 20 gauge angiocatheter.

General anesthesia will be started. A baseline glucose level will be taken from a blood gas sample, from the arterial line inserted at the beginning of the surgery.

In the Control group, patients' glucose levels will be managed as per the anesthesiologist and/or the anesthesia resident in charge of intraoperative anesthesia management of the patients. The patient will be given actrapid insulin using the glucose sliding scale for diabetic patients as set by the protocol set at AUBMC (mentioned in methodology).

The anesthesia resident will be just asked to take a blood gas sample for the patient every 30 minutes without telling him/her about the purpose of the study, so he/she will be blinded and will act accordingly (including administering insulin to the patient or just monitoring the blood glucose levels without intervening). At the end of the surgery a copy of the blood gas samples and chart of the patients will be collected.

In the Experimental group, patients will be treated using an automated protocol consisting of an insulin infusion pump named The Space Glucose Control System by B. Braun, in Melsungen, Germany. The Space Glucose Control system is a Class IIb medical device. The manufacturer, B. Braun, received the first CE mark in June 2004. The most recent renewal was in May 2013. At the bottom of this system, a central user interface is connected with a touch screen interface in order to enter the data. The glucose reading as measured has to be entered manually by the medical house staff (anesthesia resident) via the touch screen display. Based on this input the system gives advice on the insulin infusion rate. The suggested insulin infusion is displayed on the screen, but has to be entered manually and therefore confirmed by the medical staff.

For glucose measurement, a sample of blood gas will be taken every half an hour. Actrapid HM will be used in a 4IU/ ml concentration for infusion in a 50 ml syringe.

The range of glucose will be recorded throughout the intra-operative period. The number of hypoglycemic (<70mg/dl) and hyperglycemic (> 200mg/dl) events will be recorded.

Insulin allergy in patients with diabetes mellitus is a rare condition. Signs and symptoms including angioedema, hypotension, urticaria and rash, if present, are usually noticed immediately following the injection. Patients suspected of having insulin allergy will be treated by stopping the infusion, administering antihistaminic H2 and H1 blockers, corticosteroids and pressors depending on the magnitude of the allergic reaction.

Hypoglycemia defined as blood glucose level less than 70 mg/dl, will be detected and treated promptly to provide a rise in blood glucose to a safe level in order to eliminate any potential harm. The intervention will include intravenous infusion of 100 to 200 ml of D5 water over 1 to 3 minutes and repeating blood glucose level after 15 minutes to reach a target blood sugar of 100. The same intervention will be repeated in case this level wasn't reached and patient will be withdrawn from the study after two failed correction and will be treated more aggressively with an infusion of D10W.

ELIGIBILITY:
Inclusion Criteria:

* Type I or type II diabetic patients from both genders aged between 40 - 75 years, who are ASA III-IV undergoing Cardiopulmonary Bypass surgery under general anesthesia for more than 4 hours and requiring the insertion of an arterial line.

Exclusion Criteria:

* Critically ill patients ASA V
* Pregnant patients
* Patients' refusal to consent
* Emergency or lifesaving cases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who will have a serum glucose level between 140-180mg/dl during surgery. | Throughout the surgery period and postoperatively (admission to the CSU)
  The reduction of this percentage to less than 10% with the fully automated algorithm as clinically significant
Percentage of patients who had hyperglycemic events | Throughout the surgery periodThroughout the surgery period and postoperatively (admission to the CSU)
  At least one hyperglycemic event over the surgery time
Percentage of patients who had hypoglycemic events | Throughout the surgery periodThroughout the surgery period and postoperatively (admission to the CSU)
  At least one hypoglycemic event over the surgery time

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Kaddoum R, Khalili A, Shebbo FM, Ghanem N, Daher LA, Ali AB, Chehade NEH, Maroun P, Aouad MT. Automated versus conventional perioperative glycemic control in adult diabetic patients undergoing open heart surgery. BMC Anesthesiol. 2022 Jun 16;22(1):184. doi: 10.1186/s12871-022-01721-6. PMID 35710339